CLINICAL TRIAL: NCT04166084
Title: The Effect of Trunk Stabilization Exercises on Postural Stability at Lipoedema Patients
Brief Title: Trunk Stabilization Exercises at Lipoedema Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Alis Kostanoğlu, Assist. Prof., Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bvuakos1
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Lipedema
Keywords: lipedema; postural stability; trunk stabilization exercises
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients in this group will receive active ROM exercises, 10 repeats X 3 times a day, 5 days a week for 6 weeks. All exercises will be performed at home .
  Interventions: Other: Active ROM Exercises
- Training group (Experimental): I addition to active ROM exercises, patients in this group will also receive trunk stabilization exercises training for 45 minutes, 2 times a week for 6 weeks. All exercises sessions will be supervised by a physiotherapist in a clinic per week.
  Interventions: Other: Active ROM Exercises; Other: Trunk Stabilization Exercises Training

INTERVENTIONS:
Other: Active ROM Exercises — Active ROM exercises programme will include hip flexion-extention, hip abduction-adduction, hip internal-external rotation, knee flexion-extention and ankle dorsi-plantar flextion exercises.
Other: Trunk Stabilization Exercises Training — Trunk stabilization exercises training will be given under the supervision of a physiotherapist. This training exercises will include diphragmatic exrecises, posterior pelvic tilt exercises, abdominal streghtening exercises,
  Arms: Training group

SUMMARY:
Lipedema is a chronic, progressive adipose tissue disorder that is mostly seen as a symmetrical growth of the hips and legs, affecting women. The aim of this study is to investigate the effect of trunk stabilization exercises in addition to active range of motion exercises on body composition, pain, edema, trunk endurance, functional capacity and postural stability.

DETAILED DESCRIPTION:
Thirty female patients with upper and lower leg lipedemia were included in the study.

Subjects were divided into two groups as experimental (n = 15) and control (n = 15).

The physiotherapy program of the control group will consist of active range of motion exercises and the physiotherapy program in the experimental group will include active range of motion exercises as well as trunk stabilization exercises. After recording demographic data of all subjects, limb volume (environmental measurement), body composition analysis, trunk endurance, pain (Visual Analogue Scale), postural stability (Biodex Balance System®) and functional capacities (6-Minute Walk Test) will be taken.

After the six-week treatment program, all evaluations will be repeated. SPSS (SPSS 21.0) program was used for statistical analysis of the data. Significance level in all analyzes will be accepted as p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with lower or upper type lipedema
* to be able to understand Turkish
* being older than 18 years

Exclusion Criteria:

* diagnosed with vestibular disorders
* having orthopedic or neurologic co morbidities

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-15 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Extremity volume | Six weeks
  tape measurements
Body Composition | Six weeks
  fat mass; muscle mass
Extremity pain | Six weeks
  Visual Analog Scale
Endurance | Six weeks
  Abdominal endurance tests
Balance | Six weeks
  Change from baseline postural stability test score in BIODE Balance System at 6 weeks.